CLINICAL TRIAL: NCT05298111
Title: Acute Effect of Melon Manis Terengganu Peel Powder on Glycemic Response, Satiety, and Food Intake in Adults at Risk for Type 2 Diabetes
Brief Title: Acute Effect of MMT Peel Powder on Glycemic Response, Satiety, and Food Intake in Adults at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sultan Zainal Abidin (Other)
Collaborators: National University of Malaysia (Other); Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ong Ying Qian, Principal Investigator, Universiti Sultan Zainal Abidin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RCTOYQ
Record Dates: First submitted 2022-03-01; First posted 2022-03-28 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: At Risk of Type 2 Diabetes Mellitus
Keywords: Melon Manis Terengganu peel; Glycemic response; Perceived satiety; Food intake; At risk of type 2 diabetes
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: The respondents consumed Formulation 3 (A) and control (B) with study breakfast based on randomly assigned treatment sequences (AB, BA). Each visit was separated with three days washout period and lasted about 3 hour (starting around 8 am and finishing at approximately 11 am).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation 3 (Active Comparator): Formulated MMT peel powder (provide 5 g dietary fiber per day)
  Interventions: Other: Formulation 3
- Control (Placebo Comparator): Glucose
  Interventions: Other: Control

INTERVENTIONS:
Other: Formulation 3 — Respondents were consumed 36 g of Formulation 3 containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast
  Other Names: Formulated MMT peel powder
  Arms: Formulation 3
Other: Control — Respondents were consumed 4.5 g of control containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast
  Other Names: Glucose
  Arms: Control

SUMMARY:
Open-label, randomised, placebo-controlled, crossover study with two intervention arms. The study was conducted in 30 respondents and the primary objective is to show an improved glycemic response after Melon Manis Terengganu (MMT) peel powder consumption in people at risk of type 2 diabetes.

DETAILED DESCRIPTION:
The main aim of the study is to investigate the acute effect of MMT peel powder on glycemic response in people at risk of type 2 diabetes. Besides, the acute effect of MMT peel powder on perceived satiety and energy intake were explored.

ELIGIBILITY:
Inclusion Criteria:

* Modified Finnish Type 2 Diabetes Risk Assessment Tool (FINDRISC) score ≥ 4
* Capillary fasting blood glucose (FBG) < 7.0 mmol/L
* Malaysian
* Live, work or study in Kuala Nerus, Terengganu
* Both gender
* Age 18 to 59 years old
* Non-smoker
* Those taking supplement agree to undergo washout period of one week

Exclusion Criteria:

* Had clinical history of type 2 diabetes mellitus (T2DM)
* Capillary FBG ≥ 7.0 mmol/L
* Take oral antidiabetic agents
* Participate in other weight management programme or interventional research
* On a prescribed medical diet
* GI illnesses or conditions
* Allergy or sensitivity to study products
* Pregnant, currently breastfeeding, or planning to become pregnant
* On dietary restrictions
* Smoker

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Sakinah Harith, Principal Investigator — Universiti Sultan Zainal Abidin; Dr Norshazila Shahidan, Principal Investigator — Universiti Sultan Zainal Abidin; Prof Madya Dr Mohd Razif Shahril, Principal Investigator — National University of Malaysia; Prof Madya Dr Hermizi Hapidin, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Food Preparation and Therapeutic Diet Lab, Faculty of Health Sciences, Universiti Sultan Zainal Abidin, Gong Badak Campus, Kuala Terengganu, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teh CH, Lim KK, Chan YY, Lim KH, Azahadi O, Hamizatul Akmar AH, Ummi Nadiah Y, Syafinaz MS, Kee CC, Yeo PS, Fadhli Y. The prevalence of physical activity and its associated factors among Malaysian adults: findings from the National Health and Morbidity Survey 2011. Public Health. 2014 May;128(5):416-23. doi: 10.1016/j.puhe.2013.10.008. Epub 2014 Apr 13. PMID 24726414
- [Background] Tey SL, Salleh NB, Henry J, Forde CG. Effects of aspartame-, monk fruit-, stevia- and sucrose-sweetened beverages on postprandial glucose, insulin and energy intake. Int J Obes (Lond). 2017 Mar;41(3):450-457. doi: 10.1038/ijo.2016.225. Epub 2016 Dec 13. PMID 27956737
- [Derived] Ong YQ, Harith S, Shahril MR, Shahidan N, Hapidin H. Acute effect of Melon Manis Terengganu peel powder on glycemic response, perceived satiety, and food intake: a randomized, placebo-controlled crossover trial in adults at risk of type 2 diabetes. BMC Nutr. 2022 Aug 8;8(1):75. doi: 10.1186/s40795-022-00572-1. PMID 35941609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 participants were screened for eligibility between 18th August 2021 and 18th October 2021 in Kuala Nerus, Terengganu, Malaysia,
Pre-assignment Details: 36 of 120 participants were randomized. 84 participants did not meet inclusion criteria.
Groups:
- Formulation 3, Then Control: Participants first consumed 36 g of Formulated MMT peel powder containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast. After a washout period of 3 days, they then consumed 4.5 g glucose containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast.
- Control, Then Formulation 3: Participants first consumed 4.5 of glucose containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast. After a washout period of 3 days, they then consumed 36 g formulated MMT peel powder containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast.
Period: First Intervention
Arm/Group | Formulation 3, Then Control | Control, Then Formulation 3
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Washout (3 Days)
Arm/Group | Formulation 3, Then Control | Control, Then Formulation 3
Started | 18 | 18
Completed | 15 | 15
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3
Period: Second Intervention
Arm/Group | Formulation 3, Then Control | Control, Then Formulation 3
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Formulation 3 Then Control: Formulated MMT peel powder (provide 5 g dietary fiber per day)
  Respondents were consumed 36 g of Formulation 3 then 4.5 g of control, both containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast.
- Control Then Formulation 3: Glucose
  Control: Respondents were consumed 4.5 g of control then 36 g of Formulation 3, both containing 4.5 g of available carbohydrate dissolved in 180 ml water with study breakfast
- Total: Total of all reporting groups
Arm/Group | Formulation 3 Then Control | Control Then Formulation 3 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (4.5) | 37.9 (6.8) | 36.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Malaysia | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Levels
Description: Blood glucose were measured using glucometer (Accu Chek Performa, New South Wales, Australia) from finger-prick blood samples according to the standard operating procedure at baseline (0 min), 30, 60, 90 and 120 minutes.
Time Frame: Baseline (0 min), 30, 60, 90 and 120 minutes on Day 1 and Day 4 of both study visits
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
mmol/L
  0 min | 5.6 (0.4) | 5.7 (0.4)
  30 min | 6.7 (0.6) | 7.7 (0.7)
  60 min | 7.4 (1.0) | 8.2 (1.2)
  90 min | 6.9 (0.8) | 7.0 (1.0)
  120 min | 6.5 (0.6) | 6.1 (0.6)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p < 0.001, ANCOVA

2. Secondary Outcome: Perceived Satiety (Area Under the Curve)
Description: Perceived satiety measurements were rated using a 10-cm visual analogue scale (VAS) which consisted of hunger (How hungry are you?), fullness (How full are you?), desire to eat (How strong is your desire to eat?), prospective food consumption (How much would you be able to eat right now?) and thirstiness (How thirsty are you?) (Tey, Salleh, Henry, & Forde, 2017). The scale ranged from 0 (not at all) to 10 (very much) measured at baseline (0 min), 30, 60, 90 and 120 minutes. The area under the curve was calculated using trapezoid rule.
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Error); unit: score on a scale*min
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
score on a scale*min
  Hunger | 200.5 (22.3) | 277 (32.4)
  Fullness | 912 (34) | 822.5 (41.6)
  Desire to eat | 231 (21.9) | 329 (32.4)
  Prospective food consumption | 263 (31) | 344.5 (35)
  Thirstiness | 486.5 (51.5) | 499.5 (45.1)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p < 0.001, Paired t-test

3. Secondary Outcome: Food Intake
Description: The respondents were asked to record all the food or drink they had consumed including sauces, soup and gravies using household measures once they woke up in the morning until they went to sleep at night.
Time Frame: Day 1 and 4 of both study visits
Measure: Median (Full Range); unit: g
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
g
  Carbohydrate | 219.3 [163.3 to 334.5] | 225.2 [143.2 to 371.6]
  Protein | 74.1 [52.2 to 106.4] | 75.3 [55.0 to 112.3]
  Fat | 74.3 [46.7 to 108.9] | 77.2 [50.3 to 118.5]
  Dietary fiber | 10.9 [8.2 to 13.9] | 6.1 [2.7 to 10.4]
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p < 0.001, Sign test

4. Secondary Outcome: Calories Intake
Description: as for outcome 3
Time Frame: Day 1 and day 4 of both study visits
Measure: Median (Full Range); unit: kcal
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
kcal | 1796 [1424 to 2569] | 1893 [1434 to 2476]
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.001, Sign test

5. Other Pre Specified Outcome: Body Weight (kg)
Description: Body weight was taken at every study visit.
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
kg | 75.1 (14.9) | 75.1 (15.0)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.894, Paired t-test

6. Other Pre Specified Outcome: Height (cm)
Description: Height was taken at every study visit.
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
cm | 158.6 (6.3) | 158.6 (6.4)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.629, Paired t-test

7. Other Pre Specified Outcome: Body Mass Index (BMI) (kg/m^2)
Description: BMI was calculated using formula = body weight (kg)/height (m)^2
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
kg/m^2 | 29.8 (5.1) | 29.8 (5.1)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.653, Paired t-test

8. Other Pre Specified Outcome: % Body Fat
Description: % body fat was taken at every study visit.
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
Percentage | 38.9 (8.1) | 39.0 (8.3)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.624, Paired t-test

9. Other Pre Specified Outcome: Waist Circumference (cm)
Description: Waist circumference was taken at every study visit.
Time Frame: Day 1 and 4 of both study visits
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
cm | 91.2 (11.0) | 91.0 (11.3)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.414, Paired t-test

10. Other Pre Specified Outcome: Blood Pressure
Description: Blood pressure was measured using an Omron automatic digital blood pressure monitor (Omron HEM-7221) in a seated position at all visits after 5 min of sitting.
Time Frame: Day 1 and 4 of both study visits
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Formulation 3 | Control
Number analyzed (Participants) | 30 | 30
mmHg
  systolic blood pressure | 124 (14) | 122 (15)
  diastolic blood pressure | 77 (9) | 75 (9)
Statistical Analysis 1: Comparison: Formulation 3 vs Control; Test type: Superiority; p = 0.105, Paired t-test

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored or assessed.
Arm/Group | Formulation 3 | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Since this is an acute feeding study, thus the acute findings cannot translate to a long-term benefit. Next, due to limitations in budgeting, the biochemical parameters such as serum insulin, lipid profiles and appetite hormones were not assessed. Therefore, satiety was only measured using subjective means instead of assessed by physiological markers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT05298111/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT05298111/SAP_002.pdf
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT05298111/ICF_000.pdf